CLINICAL TRIAL: NCT00449657
Title: Phase II Trial of Pulsed Paclitaxel With Concurrent Radiotherapy,and Adjuvant Chemotherapy in Stage III Non-Small Cell Lung Cancer
Brief Title: Phase II Trial of Pulsed Taxol With Concurrent Thoracic Radiotherapy, & Adjuvant Chemo in Stage III NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual, change in standard of care.
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJCC 07-01
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Radiotherapy; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Taxol (paclitaxel) — paclitaxel 15mg/m2 Q am on Mon/Wed/Fri
Procedure: Radiotherapy — Off cord thoracic radiotherapy 200cGy (total dose 1000cGy). Mon/Wed/Fri: radiotherapy is delivered at least 6 hrs after chemotherapy. Tue/Thurs: radiotherapy is delivered 24 hrs or less from the paclitaxel dose the day before.
  Off-cord and off-esophagus concomitant boost radiotherapy 100 cGy (total dose 500 cGy)Mon/Wed/Fri of week 5
Drug: Carboplatin — Carboplatin AUC 5mg/min/ml, prior to Gemcitabine on Wed of weeks 8 & 9
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 at a fixed dose rate of 10mg/m2/min on Wed during week 8 & 9

SUMMARY:
This is a phase II study to evaluate the toxicity and overall survival of pulsed paclitaxel with concurrent thoracic radiotherapy, and adjuvant gemcitabine and carboplatin in stage IIIA and IIIB non-small cell lung cancer

DETAILED DESCRIPTION:
OBJECTIVES Primary

1. Overall survival
2. Tumor response using RECIST criteria

Secondary

1. Determine the toxicity of the proposed treatment in this patient population.
2. Progression free survival
3. Locoregional control
4. Distant failure

STUDY DESIGN

Description of the Study Phase II study to evaluate the toxicity and overall survival of pulsed paclitaxel with concurrent thoracic radiotherapy, and adjuvant gemcitabine and carboplatin in stage IIIA and IIIB non-small cell lung cancer.

Rationale for Study Design The proposed doses of gemcitabine, carboplatin, paclitaxel, and thoracic radiation therapy have been previously studied and deemed safe. The design of this study is not to find the maximum tolerated dose (MTD) of these agents, but to study the toxicity and overall survival from this combination.

Outcome Measures Primary Outcome Measures

1. Overall survival
2. Tumor response using RECIST criteria

Secondary Outcome Measures

1. Locoregional control
2. Distant Failure
3. Progression free survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have: IIIA or IIIB non-small cell lung cancer by radiographic or surgical staging, excluding: superior sulcus tumors, tumors with associated atelectasis or obstructive pneumonitis of the entire lung, and tumors with a malignant pleural effusion.
2. Patients will be included in the study based on the following criteria:

   * Patients must be older than 18 years old.
   * Patients must have a Zubrod performance status of 0 to 2
   * Patients with adequate bone marrow function
   * Patients with adequate renal function
   * Patients with adequate hepatic function
   * Patients of childbearing potential must have a negative serum pregnancy test and use an effective form of contraception.
   * Patients who are suitable for treatment with radical intent using concurrent chemotherapy and radiation.
   * Patients who have signed an approved informed consent and authorization permitting release of personal health information.

Exclusion Criteria:

1. Disease-Specific Exclusions

   * Superior sulcus tumors
   * Atelectasis or obstructive pneumonitis of the entire lung
   * Malignant pleural effusion
2. General Medical Exclusions

   * Surgical candidates
   * Patients who are pregnant at the time of diagnosis
   * Serious concomitant systemic disorders incompatible with the study
   * Inability to comply with study and/or follow-up procedures
   * Life expectancy of less than 12 weeks
   * Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
   * Patients with septicemia or severe infection.
   * Patients who have circumstances that will not permit completion of this study or the required follow-up
   * Patients with any contraindication to gemcitabine, carboplatin, or paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Tumor response using RECIST criteria | 12/31/2014

SECONDARY OUTCOMES:
Locoregional control | 12/31/2014
Distant failure | 12/31/2014
Progression free survival | 12/31/2014

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walker, MD, Principal Investigator — Brody School of Medicine at East Carolina University
Locations (1):
- Brody School of Medicine at East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Background] Travis WD, Lubin J, Ries L, Devesa S. United States lung carcinoma incidence trends: declining for most histologic types among males, increasing among females. Cancer. 1996 Jun 15;77(12):2464-70. doi: 10.1002/(SICI)1097-0142(19960615)77:123.0.CO;2-M. PMID 8640694
- [Background] Pisani P, Parkin DM, Ferlay J. Estimates of the worldwide mortality from eighteen major cancers in 1985. Implications for prevention and projections of future burden. Int J Cancer. 1993 Dec 2;55(6):891-903. doi: 10.1002/ijc.2910550604. PMID 8253525
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Peto R, Lopez AD, Boreham J, Thun M, Heath C Jr. Mortality from tobacco in developed countries: indirect estimation from national vital statistics. Lancet. 1992 May 23;339(8804):1268-78. doi: 10.1016/0140-6736(92)91600-d. PMID 1349675
- [Background] Hoffman PC, Mauer AM, Vokes EE. Lung cancer. Lancet. 2000 Feb 5;355(9202):479-85. doi: 10.1016/S0140-6736(00)82038-3. PMID 10841143
- [Background] Jemal A, Murray T, Samuels A, Ghafoor A, Ward E, Thun MJ. Cancer statistics, 2003. CA Cancer J Clin. 2003 Jan-Feb;53(1):5-26. doi: 10.3322/canjclin.53.1.5. PMID 12568441
- [Background] Onishi H, Araki T, Shirato H, Nagata Y, Hiraoka M, Gomi K, Yamashita T, Niibe Y, Karasawa K, Hayakawa K, Takai Y, Kimura T, Hirokawa Y, Takeda A, Ouchi A, Hareyama M, Kokubo M, Hara R, Itami J, Yamada K. Stereotactic hypofractionated high-dose irradiation for stage I nonsmall cell lung carcinoma: clinical outcomes in 245 subjects in a Japanese multiinstitutional study. Cancer. 2004 Oct 1;101(7):1623-31. doi: 10.1002/cncr.20539. PMID 15378503
- [Background] Chen Y, Pandya K, Keng PC, Johnstone D, Li J, Lee YJ, Smudzin T, Okunieff P. Phase I/II clinical study of pulsed paclitaxel radiosensitization for thoracic malignancy: a therapeutic approach on the basis of preclinical research of human cancer cell lines. Clin Cancer Res. 2003 Mar;9(3):969-75. PMID 12631594
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Hotta K, Matsuo K, Ueoka H, Kiura K, Tabata M, Tanimoto M. Meta-analysis of randomized clinical trials comparing Cisplatin to Carboplatin in patients with advanced non-small-cell lung cancer. J Clin Oncol. 2004 Oct 1;22(19):3852-9. doi: 10.1200/JCO.2004.02.109. Epub 2004 Aug 23. PMID 15326195
- [Background] Zatloukal P, Petruzelka L, Zemanova M, Kolek V, Skrickova J, Pesek M, Fojtu H, Grygarkova I, Sixtova D, Roubec J, Horenkova E, Havel L, Prusa P, Novakova L, Skacel T, Kuta M. Gemcitabine plus cisplatin vs. gemcitabine plus carboplatin in stage IIIb and IV non-small cell lung cancer: a phase III randomized trial. Lung Cancer. 2003 Sep;41(3):321-31. doi: 10.1016/s0169-5002(03)00233-2. PMID 12928123
- [Background] Bajetta E, Stani SC, De Candis D, Zaffaroni N, Zilembo N, Cortinovis D, Aglione S, Mariani L, Formisano B, Bidoli P. Preclinical and clinical evaluation of four gemcitabine plus carboplatin schedules as front-line treatment for stage IV non-small-cell lung cancer. Ann Oncol. 2003 Feb;14(2):242-7. doi: 10.1093/annonc/mdg060. PMID 12562651
- [Background] Grunewald R, Kantarjian H, Keating MJ, Abbruzzese J, Tarassoff P, Plunkett W. Pharmacologically directed design of the dose rate and schedule of 2',2'-difluorodeoxycytidine (Gemcitabine) administration in leukemia. Cancer Res. 1990 Nov 1;50(21):6823-6. PMID 2208147
- [Background] Abbruzzese JL, Grunewald R, Weeks EA, Gravel D, Adams T, Nowak B, Mineishi S, Tarassoff P, Satterlee W, Raber MN, et al. A phase I clinical, plasma, and cellular pharmacology study of gemcitabine. J Clin Oncol. 1991 Mar;9(3):491-8. doi: 10.1200/JCO.1991.9.3.491. PMID 1999720
- [Background] Soo RA, Wang LZ, Tham LS, Yong WP, Boyer M, Lim HL, Lee HS, Millward M, Liang S, Beale P, Lee SC, Goh BC. A multicentre randomised phase II study of carboplatin in combination with gemcitabine at standard rate or fixed dose rate infusion in patients with advanced stage non-small-cell lung cancer. Ann Oncol. 2006 Jul;17(7):1128-33. doi: 10.1093/annonc/mdl084. Epub 2006 May 2. PMID 16670205
- [Derived] Zhang J, Gay HA, Russo S, Parent T, Aljumaily R, Walker PR. Phase II study of low-dose paclitaxel with timed thoracic radiotherapy followed by adjuvant gemcitabine and carboplatin in unresectable stage III non-small cell lung cancer. Lung Cancer. 2014 Jan;83(1):67-72. doi: 10.1016/j.lungcan.2013.09.007. Epub 2013 Sep 25. PMID 24246506